CLINICAL TRIAL: NCT01301079
Title: Evaluation of the Effect of Ketamine on Remifentanil-induced Hyperalgesia Using Filaments, an Algometer, and Interleukins: a Double-blind, Randomized Study
Brief Title: Evaluation of the Effect of Ketamine on Remifentanil-induced Hyperalgesia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Plínio da Cunha Leal, Master's degree, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: anaana
Record Dates: First submitted 2011-02-22; First posted 2011-02-23 (Estimated); Results first posted 2014-11-10 (Estimated); Last update posted 2014-11-10 (Estimated); Status verified 2014-10

CONDITIONS: Pain; Hyperalgesia; Inflammatory Response
Keywords: Remifentanil; Hyperalgesia; Ketamine; Von Frey's filament; Algometer; Interleukines; Opioid-induced hyperalgesia
MeSH Terms: conditions — Pain; Hyperalgesia | interventions — Ketamine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ketamine (Active Comparator): A cardioscope, a capnograph, a pulse oximeter, and a noninvasive blood pressure meter were used to monitor the patients. Propofol (2-4 mg/kg), remifentanil (1 μg/kg), and atracurium (0.5 mg/kg) were administered for intubation. Atracurium was titrated to maintain muscle relaxation. Anesthesia was maintained with remifentanil, 0.8% isoflurane, and 50% oxygen without nitrous oxide. Infusion of the solutions was continued until skin closure.
  The patients in group ketamine received remifentanil (0.4 μg/kg/min) and ketamine (5 μg/kg/min).
  Remifentanil was administered as necessary until skin closure. Neostigmine was used for antagonizing the neuromuscular block.
  Interventions: Drug: Ketamine
- Saline (Placebo Comparator): A cardioscope, a capnograph, a pulse oximeter, and a noninvasive blood pressure meter were used to monitor the patients. Propofol (2-4 mg/kg), 1 μg/kg remifentanil, and atracurium (0.5 mg/kg) were administered for intubation. Atracurium was titrated to maintain muscle relaxation. Anesthesia was maintained with remifentanil, 0.8% isoflurane, and 50% oxygen without nitrous oxide. Infusion of the solutions was continued until skin closure.
  The patients in group saline received remifentanil (0.4 μg/kg/min) and saline solution.
  Remifentanil was administered as necessary until skin closure. Neostigmine was used for antagonizing the neuromuscular block.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Ketamine — Patients in group ketamine was administrated ketamine (5mcg/kg/min) during the surgery.
  Arms: Ketamine
Drug: Saline — Patients in group N (placebo) was administrated saline during surgery.
  Arms: Saline

SUMMARY:
The aim of this study was to determine if the addition of ketamine reduces remifentanil-induced hyperalgesia, improves its analgesic effect, inhibits IL(interleukin)-6 and IL-8 (inflammatory cytokines), and stimulates IL-10 (an anti-inflammatory cytokine).

DETAILED DESCRIPTION:
Opioids are very effective in pain relief, but they might lower pain threshold, making the patient more sensitive to a pain stimulus, a condition known as hyperalgesia [Angst; Clarck, 2006]. Opioid-induced hyperalgesia (OIH) is usually defined as a reduction in nociceptive thresholds in the peripheral field of the sensitized fibers [Koppert et al., 2003], and it is associated with increased pain and higher demand for postoperative analgesia [Guignard et al., 2000]. This phenomenon adversely impacts pain control, and has been suggested to occur in the peri-operative context, especially associated with the use of remifentanil, a short-acting opioid [Guignard et al., 2000].

Several mechanisms have been proposed to explain the hyperalgesia phenomenon, but the most important seems to be the activation of N-methyl-D-aspartate (NMDA) receptors [Célèrier et al., 2000]. Ketamine is a NMDA receptor antagonist that has been shown to reduce postoperative pain and the need for postoperative anesthetics and analgesics. Therefore, it is proposed that ketamine could prevent hyperalgesia, resulting in more effective and long-lasting postsurgical analgesia [Célèrier et al. 2000].

The results of studies of low dose of ketamine in the prevention of remifentanil-induced hyperalgesia are controversial. Joly et al. [2005] demonstrated a reduction in the consumption of opioids and in hyperalgesia assessed with monofilaments. However, Engelhardt et al [2008] showed no differences in pain scores or in postoperative opioid consumption.

In addition, some authors observed higher levels of proinflammatory cytokines, associated with increased pain in mice receiving chronic opioid (morphine) infusion [Johnston et al., 2004; Liang et al., 2008]. Also, administration of proinflammatory cytokine inhibitors reduced phosphorylation of NMDA receptors [Zhang et al., 2008]. However, no study has examined the relationship between the use of remifentanil, the most frequently implicated opioid in OIH [Guignard et al., 2000], ketamine (drug capable of inhibiting NMDA-receptors and cytokines) [Dale et al., 2012], and the inflammatory response.

The aim of this study was to determine if the addition of ketamine reduces remifentanil-induced hyperalgesia, improves its analgesic effect, inhibits IL-6 and IL-8 (inflammatory cytokines), and stimulates IL-10 (an anti-inflammatory cytokine) in patients submitted to laparoscopic cholecystectomy, a procedure with an usually neglected potential for postoperative pain and that has been poorly investigated in association with OIH.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* both sexes
* ASA physical status I or II
* undergoing laparoscopic cholecystectomy

Exclusion Criteria:

* chronic users of analgesics or had used opioids within 12 h of surgery
* history of drug or alcohol abuse or psychiatric disorder
* contraindications to self-administration of opioids (ie, unable to understand the patient-controlled analgesia [PCA] device)
* contraindication for the use of ketamine, such as a psychiatric disorder, acute cardiovascular disorder, or unstable hypertension

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-09; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Plínio da Cunha Leal, PhD, Principal Investigator — Federal University of São Paulo
Locations (1):
- Federal University of São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Liang D, Shi X, Qiao Y, Angst MS, Yeomans DC, Clark JD. Chronic morphine administration enhances nociceptive sensitivity and local cytokine production after incision. Mol Pain. 2008 Feb 22;4:7. doi: 10.1186/1744-8069-4-7. PMID 18294378
- [Background] Zhang RX, Li A, Liu B, Wang L, Ren K, Zhang H, Berman BM, Lao L. IL-1ra alleviates inflammatory hyperalgesia through preventing phosphorylation of NMDA receptor NR-1 subunit in rats. Pain. 2008 Apr;135(3):232-239. doi: 10.1016/j.pain.2007.05.023. Epub 2007 Aug 6. PMID 17689191
- [Background] Dale O, Somogyi AA, Li Y, Sullivan T, Shavit Y. Does intraoperative ketamine attenuate inflammatory reactivity following surgery? A systematic review and meta-analysis. Anesth Analg. 2012 Oct;115(4):934-43. doi: 10.1213/ANE.0b013e3182662e30. Epub 2012 Jul 23. PMID 22826531
- [Result] Angst MS, Clark JD. Opioid-induced hyperalgesia: a qualitative systematic review. Anesthesiology. 2006 Mar;104(3):570-87. doi: 10.1097/00000542-200603000-00025. PMID 16508405
- [Result] Koppert W, Sittl R, Scheuber K, Alsheimer M, Schmelz M, Schuttler J. Differential modulation of remifentanil-induced analgesia and postinfusion hyperalgesia by S-ketamine and clonidine in humans. Anesthesiology. 2003 Jul;99(1):152-9. doi: 10.1097/00000542-200307000-00025. PMID 12826855
- [Result] Guignard B, Bossard AE, Coste C, Sessler DI, Lebrault C, Alfonsi P, Fletcher D, Chauvin M. Acute opioid tolerance: intraoperative remifentanil increases postoperative pain and morphine requirement. Anesthesiology. 2000 Aug;93(2):409-17. doi: 10.1097/00000542-200008000-00019. PMID 10910490
- [Result] Celerier E, Rivat C, Jun Y, Laulin JP, Larcher A, Reynier P, Simonnet G. Long-lasting hyperalgesia induced by fentanyl in rats: preventive effect of ketamine. Anesthesiology. 2000 Feb;92(2):465-72. doi: 10.1097/00000542-200002000-00029. PMID 10691234
- [Result] Joly V, Richebe P, Guignard B, Fletcher D, Maurette P, Sessler DI, Chauvin M. Remifentanil-induced postoperative hyperalgesia and its prevention with small-dose ketamine. Anesthesiology. 2005 Jul;103(1):147-55. doi: 10.1097/00000542-200507000-00022. PMID 15983467
- [Result] Engelhardt T, Zaarour C, Naser B, Pehora C, de Ruiter J, Howard A, Crawford MW. Intraoperative low-dose ketamine does not prevent a remifentanil-induced increase in morphine requirement after pediatric scoliosis surgery. Anesth Analg. 2008 Oct;107(4):1170-5. doi: 10.1213/ane.0b013e318183919e. PMID 18806023
- [Result] Johnston IN, Milligan ED, Wieseler-Frank J, Frank MG, Zapata V, Campisi J, Langer S, Martin D, Green P, Fleshner M, Leinwand L, Maier SF, Watkins LR. A role for proinflammatory cytokines and fractalkine in analgesia, tolerance, and subsequent pain facilitation induced by chronic intrathecal morphine. J Neurosci. 2004 Aug 18;24(33):7353-65. doi: 10.1523/JNEUROSCI.1850-04.2004. PMID 15317861

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Inclusion criteria were: ≥18 years of age, any gender, classified as American Society of Anesthesiologists (ASA) Physical Status I or II, and undergoing laparoscopic cholecystectomy at Hospital São Paulo/Federal University of São Paulo, from September 2010 to September 2012.
Groups:
- Ketamine: A cardioscope, a capnograph, a pulse oximeter, and a noninvasive blood pressure meter were used to monitor the patients. Propofol (2-4 mg/kg), 1 μg/kg remifentanil, and atracurium (0.5 mg/kg) were administered for intubation. Atracurium was titrated to maintain muscle relaxation. Anesthesia was maintained with remifentanil, 0.8% isoflurane, and 50% oxygen without nitrous oxide. Infusion of the solutions was continued until skin closure.
  The patients in group ketamine received remifentanil (0.4 μg/kg/min) and ketamine (5 μg/kg/min). Neostigmine was used for antagonizing the neuromuscular block.
Period: Overall Study
Arm/Group | Ketamine | Saline
Started | 30 | 30
Completed | 28 | 28
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Ketamine: A cardioscope, a capnograph, a pulse oximeter, and a noninvasive blood pressure meter were used to monitor the patients. Propofol (2-4 mg/kg), 1 μg/kg remifentanil, and atracurium (0.5 mg/kg) were administered for intubation. Atracurium was titrated to maintain muscle relaxation. Anesthesia was maintained with remifentanil, 0.8% isoflurane, and 50% oxygen without nitrous oxide. Infusion of the solutions was continued until skin closure. The patients in group 1 (G1) received remifentanil (0.4 μg/kg/min) and ketamine (5 μg/kg/min).
  Ketamine : Patients in group ketamine will receive ketamine (5mcg/kg/min) during the surgery.
- Saline: A cardioscope, a capnograph, a pulse oximeter, and a noninvasive blood pressure meter were used to monitor the patients. Propofol (2-4 mg/kg), 1 μg/kg remifentanil, and atracurium (0.5 mg/kg) were administered for intubation. Atracurium was titrated to maintain muscle relaxation. Anesthesia was maintained with remifentanil, 0.8% isoflurane, and 50% oxygen without nitrous oxide. Infusion of the solutions was continued until skin closure. Patients in group 2 (G2) received remifentanil (0.4 μg/kg/min) and saline solution.
  Saline : Patients in group N (placebo)will receive saline during surgery.
- Total: Total of all reporting groups
Arm/Group | Ketamine | Saline | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 28 | 57
  >=65 years | 1 | 2 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.80 (13.10) | 43.40 (15.90) | 44.60 (14.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 24 | 49
  Male | 5 | 6 | 11
Region of Enrollment [Number; unit: participants]
  Brazil | 30 | 30 | 60

OUTCOME MEASURES:

1. Secondary Outcome: Time to First Morphine Supplementation
Time Frame: 24 hours
Measure: Median (Full Range); unit: minutes
Groups:
- Ketamine: A cardioscope, a capnograph, a pulse oximeter, and a noninvasive blood pressure meter were used to monitor the patients. Propofol (2-4 mg/kg), 1 μg/kg remifentanil, and atracurium (0.5 mg/kg) were administered for intubation. Atracurium was titrated to maintain muscle relaxation. Anesthesia was maintained with remifentanil, 0.8% isoflurane, and 50% oxygen without nitrous oxide. Infusion of the solutions was continued until skin closure.
  The patients in group ketamine received remifentanil (0.4 μg/kg/min) and ketamine (5 μg/kg/min). Remifentanil was administered as necessary until skin closure. Neostigmine was used for antagonizing the neuromuscular block.
Arm/Group | Ketamine | Saline
Number analyzed (Participants) | 28 | 28
minutes | 18 [0 to 600] | 15 [2 to 130]
Statistical Analysis 1: Comparison: Ketamine vs Saline; Test type: Superiority or Other; p = 0.113, Mann-Whitney

2. Secondary Outcome: Morphine Consumption Within 24 h
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: milligram
Arm/Group | Ketamine | Saline
Number analyzed (Participants) | 28 | 28
milligram | 27.40 (18.30) | 27.70 (12.90)
Statistical Analysis 1: Comparison: Ketamine vs Saline; Test type: Superiority or Other; p = 0.946, t-test, 2 sided

3. Secondary Outcome: Hyperalgesia in the Preoperative Period as Measured With Monofilaments in Thenar Eminence
Description: The pain threshold was assessed using six von Frey monofilaments (0,05 g; 0,2 g; 2 g; 4 g; 10 g e 300 g) in thenar eminence in the preoperative period. The use of different von Frey monofilaments, starting with the lightest and ending with the heaviest, was separated by at least 30 seconds to reduce any anticipated responses due to a new stimulation that was performed too soon after the preceding stimulation. Three assessments were made for each monofilament, and this was considered positive when the patient responded to two of the determinations for each monofilament.
Time Frame: Before the procedure (Baseline)
Measure: Mean (Standard Deviation); unit: gram
Arm/Group | Ketamine | Saline
Number analyzed (Participants) | 28 | 28
gram | 300 (0) | 300 (0)
Statistical Analysis 1: Comparison: Ketamine vs Saline; Test type: Superiority or Other; p = 0.999, t-test, 2 sided

4. Secondary Outcome: Hyperalgesia in the Postoperative Period as Measured With Monofilaments in Thenar Eminence
Description: The pain threshold was assessed using six von Frey monofilaments (0,05 g; 0,2 g; 2 g; 4 g; 10 g e 300 g) in thenar eminence in the postoperative period (24 hours after procedure). The use of different von Frey monofilaments, starting with the lightest and ending with the heaviest, was separated by at least 30 seconds to reduce any anticipated responses due to a new stimulation that was performed too soon after the preceding stimulation. Three assessments were made for each monofilament, and this was considered positive when the patient responded to two of the determinations for each monofilament.
Time Frame: 24 hours after procedure
Measure: Mean (Standard Deviation); unit: gram
Groups:
- Ketamine: A cardioscope, a capnograph, a pulse oximeter, and a noninvasive blood pressure meter were used to monitor the patients. Propofol (2-4 mg/kg), 1 μg/kg remifentanil, and atracurium (0.5 mg/kg) were administered for intubation. Atracurium was titrated to maintain muscle relaxation. Anesthesia was maintained with remifentanil, 0.8% isoflurane, and 50% oxygen without nitrous oxide. Infusion of the solutions was continued until skin closure.
  The patients in group ketamine received remifentanil (0.4 μg/kg/min) and ketamine (5 μg/kg/min).
  Remifentanil was administered as necessary until skin closure. Neostigmine was used for antagonizing the neuromuscular block.
  Ketamine: Patients in group ketamine was administrated ketamine (5mcg/kg/min) during the surgery.
- Saline: A cardioscope, a capnograph, a pulse oximeter, and a noninvasive blood pressure meter were used to monitor the patients. Propofol (2-4 mg/kg), 1 μg/kg remifentanil, and atracurium (0.5 mg/kg) were administered for intubation. Atracurium was titrated to maintain muscle relaxation. Anesthesia was maintained with remifentanil, 0.8% isoflurane, and 50% oxygen without nitrous oxide. Infusion of the solutions was continued until skin closure.
  The patients in group saline received remifentanil (0.4 μg/kg/min) and saline solution.
  Remifentanil was administered as necessary until skin closure. Neostigmine was used for antagonizing the neuromuscular block.
  Saline: Patients in group N (placebo) was administrated saline during surgery.
Arm/Group | Ketamine | Saline
Number analyzed (Participants) | 28 | 28
gram | 290 (54.8) | 247 (115)
Statistical Analysis 1: Comparison: Ketamine vs Saline; Test type: Superiority or Other; p = 0.019, t-test, 2 sided

5. Secondary Outcome: Hyperalgesia in the Preoperative Period as Measured With Monofilaments in the Periumbilical Region
Description: The pain threshold was assessed using six von Frey monofilaments (0,05 g; 0,2 g; 2 g; 4 g; 10 g e 300 g) in the periumbilical region in the preoperative period. The use of different von Frey monofilaments, starting with the lightest and ending with the heaviest, was separated by at least 30 seconds to reduce any anticipated responses due to a new stimulation that was performed too soon after the preceding stimulation. Three assessments were made for each monofilament, and this was considered positive when the patient responded to two of the determinations for each monofilament.
Time Frame: Before the procedure (Baseline)
Measure: Mean (Standard Deviation); unit: gram
Arm/Group | Ketamine | Saline
Number analyzed (Participants) | 28 | 28
gram | 279 (77.1) | 269 (92)
Statistical Analysis 1: Comparison: Ketamine vs Saline; Test type: Superiority or Other; p = 0.652, t-test, 2 sided

6. Secondary Outcome: Hyperalgesia in the Postoperative Period as Measured With Monofilaments in the Periumbilical Region
Description: The pain threshold was assessed using six von Frey monofilaments (0,05 g; 0,2 g; 2 g; 4 g; 10 g e 300 g) in the periumbilical region in the postoperative period (24h after the procedure). The use of different von Frey monofilaments, starting with the lightest and ending with the heaviest, was separated by at least 30 seconds to reduce any anticipated responses due to a new stimulation that was performed too soon after the preceding stimulation. Three assessments were made for each monofilament, and this was considered positive when the patient responded to two of the determinations for each monofilament.
Time Frame: 24h after the procedure
Measure: Mean (Standard Deviation); unit: gram
Arm/Group | Ketamine | Saline
Number analyzed (Participants) | 28 | 28
gram | 248 (114) | 205 (140)
Statistical Analysis 1: Comparison: Ketamine vs Saline; Test type: Superiority or Other; p = 0.221, t-test, 2 sided

7. Secondary Outcome: Hyperalgesia in the Preoperative Period as Measured With Algometer in Thenar Eminence
Description: The mechanical pain threshold was evaluated using an algometer. The pressure was increased by 0.1 kgf/second until the patient complained of pain. The mean of three determinations was calculated.
Time Frame: Baseline (before the procedure)
Measure: Mean (Standard Deviation); unit: kilogram force/second
Arm/Group | Ketamine | Saline
Number analyzed (Participants) | 28 | 28
kilogram force/second | 2.51 (1.43) | 2.19 (0.92)
Statistical Analysis 1: Comparison: Ketamine vs Saline; Test type: Superiority or Other; p = 0.325, t-test, 2 sided

8. Primary Outcome: Pain 30 Minutes
Description: The scale measure pain after 30 minutes (0 - without pain and 10 worst pain possible). The individual can choose any number between 0 - 10.
Time Frame: 30 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketamine | Saline
Number analyzed (Participants) | 28 | 28
units on a scale | 5.5 (3.5) | 6.2 (2.6)
Statistical Analysis 1: Comparison: Ketamine vs Saline; Test type: Superiority or Other; p = 0.386, t-test, 2 sided

9. Primary Outcome: Pain 60 Minutes
Description: The scale measure pain after 60 minutes (0 - without pain and 10 worst pain possible). The individual can choose any number between 0 - 10.
Time Frame: 60 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Ketamine: A cardioscope, a capnograph, a pulse oximeter, and a noninvasive blood pressure meter were used to monitor the patients. Propofol (2-4 mg/kg), 1 μg/kg remifentanil, and atracurium (0.5 mg/kg) were administered for intubation. Atracurium was titrated to maintain muscle relaxation. Anesthesia was maintained with remifentanil, 0.8% isoflurane, and 50% oxygen without nitrous oxide. Infusion of the solutions was continued until skin closure.
  The patients in group 1 (G1) received remifentanil (0.4 μg/kg/min) and ketamine (5 μg/kg/min). Remifentanil was administered as necessary until skin closure. Neostigmine was used for antagonizing the neuromuscular block.
Arm/Group | Ketamine | Saline
Number analyzed (Participants) | 28 | 28
units on a scale | 4.6 (3.0) | 5.1 (2.5)
Statistical Analysis 1: Comparison: Ketamine vs Saline; Test type: Superiority or Other; p = 0.499, t-test, 1 sided

10. Primary Outcome: Pain 90 Minutes
Description: The scale measure pain after 90 minutes (0 - without pain and 10 worst pain possible). The individual can choose any number between 0 - 10.
Time Frame: 90 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketamine | Saline
Number analyzed (Participants) | 28 | 28
units on a scale | 3.4 (2.4) | 3.4 (2.3)
Statistical Analysis 1: Comparison: Ketamine vs Saline; Test type: Superiority or Other; p = 0.909, t-test, 2 sided

11. Primary Outcome: Pain 120 Minutes
Description: The scale measure pain after 120 minutes (0 - without pain and 10 worst pain possible). The individual can choose any number between 0 - 10.
Time Frame: 120 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketamine | Saline
Number analyzed (Participants) | 28 | 28
units on a scale | 2.2 (2.1) | 2.0 (1.8)
Statistical Analysis 1: Comparison: Ketamine vs Saline; Test type: Superiority or Other; p = 0.737, t-test, 2 sided

12. Primary Outcome: Pain 150 Minutes
Description: The scale measure pain after 150 minutes (0 - without pain and 10 worst pain possible). The individual can choose any number between 0 - 10.
Time Frame: 150 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketamine | Saline
Number analyzed (Participants) | 28 | 28
units on a scale | 1.4 (1.7) | 1.4 (1.6)
Statistical Analysis 1: Comparison: Ketamine vs Saline; Test type: Superiority or Other; p < 0.872, t-test, 2 sided

13. Primary Outcome: Pain 180 Minutes
Description: The scale measure pain after 180 minutes (0 - without pain and 10 worst pain possible). The individual can choose any number between 0 - 10.
Time Frame: 180 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketamine | Saline
Number analyzed (Participants) | 28 | 28
units on a scale | 1.1 (1.5) | 1.3 (1.5)
Statistical Analysis 1: Comparison: Ketamine vs Saline; Test type: Superiority or Other; p = 0.598, t-test, 2 sided

14. Primary Outcome: Pain 210 Minutes
Description: The scale measure pain after 210 minutes (0 - without pain and 10 worst pain possible). The individual can choose any number between 0 - 10.
Time Frame: 210 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketamine | Saline
Number analyzed (Participants) | 28 | 28
units on a scale | 0.9 (1.6) | 1.2 (1.5)
Statistical Analysis 1: Comparison: Ketamine vs Saline; Test type: Superiority or Other; p = 0.485, t-test, 2 sided; Mean Difference (Final Values) = 2.0

15. Primary Outcome: Pain 240 Minutes
Description: The scale measure pain after 240 minutes (0 - without pain and 10 worst pain possible). The individual can choose any number between 0 - 10.
Time Frame: 240 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketamine | Saline
Number analyzed (Participants) | 28 | 28
units on a scale | 1.0 (1.7) | 1.1 (1.5)
Statistical Analysis 1: Comparison: Ketamine vs Saline; Test type: Superiority or Other; p = 0.744, t-test, 2 sided

16. Primary Outcome: Pain 6 Hours
Description: The scale measure pain after 6 hours (0 - without pain and 10 worst pain possible). The individual can choose any number between 0 - 10.
Time Frame: 6 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketamine | Saline
Number analyzed (Participants) | 28 | 28
units on a scale | 0.9 (1.2) | 0.7 (1.0)
Statistical Analysis 1: Comparison: Ketamine vs Saline; Test type: Superiority or Other; p = 0.540, t-test, 2 sided

17. Primary Outcome: Pain 12 Hours
Description: The scale measure pain after 12 hours (0 - without pain and 10 worst pain possible). The individual can choose any number between 0 - 10.
Time Frame: 12 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketamine | Saline
Number analyzed (Participants) | 28 | 28
units on a scale | 1.6 (1.8) | 1.4 (2.0)
Statistical Analysis 1: Comparison: Ketamine vs Saline; Test type: Superiority or Other; p = 0.673, t-test, 2 sided

18. Primary Outcome: Pain 18 Hours
Description: The scale measure pain after 18 hours (0 - without pain and 10 worst pain possible). The individual can choose any number between 0 - 10.
Time Frame: 18 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketamine | Saline
Number analyzed (Participants) | 28 | 28
units on a scale | 1.5 (1.8) | 1.3 (1.6)
Statistical Analysis 1: Comparison: Ketamine vs Saline; Test type: Superiority or Other; p = 0.586, t-test, 2 sided

19. Primary Outcome: Pain 24 Hours
Description: The scale measure pain after 24 hours (0 - without pain and 10 worst pain possible). The individual can choose any number between 0 - 10.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketamine | Saline
Number analyzed (Participants) | 28 | 28
units on a scale | 1.4 (1.5) | 0.8 (1.0)
Statistical Analysis 1: Comparison: Ketamine vs Saline; Test type: Superiority or Other; p = 0.077, t-test, 2 sided

20. Secondary Outcome: Hyperalgesia in the Postoperative Period as Measured With Algometer in Thenar Eminence
Description: as for outcome 7
Time Frame: 24 h after the procedure
Measure: Mean (Standard Deviation); unit: kilogram force/second
Arm/Group | Ketamine | Saline
Number analyzed (Participants) | 28 | 28
kilogram force/second | 0.56 (0.44) | 0.51 (0.44)
Statistical Analysis 1: Comparison: Ketamine vs Saline; Test type: Superiority or Other; p = 0.677, t-test, 2 sided

21. Secondary Outcome: Hyperalgesia in the Preoperative Period as Measured With Algometer in the Periumbilical Region
Description: as for outcome 7
Time Frame: Baseline (before the surgery)
Measure: Mean (Standard Deviation); unit: kilogram force/second
Arm/Group | Ketamine | Saline
Number analyzed (Participants) | 28 | 28
kilogram force/second | 3.6 (1.5) | 3.9 (1.4)
Statistical Analysis 1: Comparison: Ketamine vs Saline; Test type: Superiority or Other; p = 0.545, t-test, 2 sided

22. Secondary Outcome: Hyperalgesia in the Postoperative Period as Measured With Algometer in the Periumbilical Region
Description: as for outcome 7
Time Frame: 24 h after the procedure
Measure: Mean (Standard Deviation); unit: kilogram force/second
Arm/Group | Ketamine | Saline
Number analyzed (Participants) | 28 | 28
kilogram force/second | 3.5 (1.6) | 3.7 (1.7)
Statistical Analysis 1: Comparison: Ketamine vs Saline; Test type: Superiority or Other; p = 0.650, t-test, 2 sided

23. Secondary Outcome: Extension of Hyperalgesia
Description: The 300-g filament was used 24 hours after the operation to induce a stimulus and delineate the extent of hyperalgesia from the periumbilical region. The stimulus was started outside the periumbilical region, where no pain sensation was reported, and continued every 0.5 cm until the 4 points of the periumbilical scar were reached (top, right side, left side, and bottom). The first point where the patient complained of pain was marked. If no pain sensation was reported, the stimulus was terminated 0.5 cm from the incision. The distance of each point from the surgical incision was measured, and the sum of the distances of the points was determined.
Time Frame: 24 hours after the procedure
Measure: Mean (Standard Deviation); unit: centimeter
Arm/Group | Ketamine | Saline
Number analyzed (Participants) | 28 | 28
centimeter | 10.61 (8.63) | 11.82 (8.36)
Statistical Analysis 1: Comparison: Ketamine vs Saline; Test type: Superiority or Other; p = 0.593, t-test, 2 sided

24. Secondary Outcome: Allodynia as Detected With a Soft Brush in the Periumbilical Region Before the Procedure
Description: The evaluations using the soft brush were performed 2-3 cm from the incision in the periumbilical region (where the large trocar was placed) before the procedure
Time Frame: Before the procedure (Baseline)
Measure: Number; unit: participants
Arm/Group | Ketamine | Saline
Number analyzed (Participants) | 28 | 28
participants | 1 | 0
Statistical Analysis 1: Comparison: Ketamine vs Saline; Test type: Superiority or Other; p = 0.313, Chi-squared

25. Secondary Outcome: Allodynia as Detected With a Soft Brush in the Periumbilical Region 24 h After the Procedure
Description: The evaluations using the soft brush were performed 2-3 cm from the incision in the periumbilical region (where the large trocar was placed) 24 h after the procedure
Time Frame: 24 h after the procedure
Measure: Number; unit: participants
Arm/Group | Ketamine | Saline
Number analyzed (Participants) | 28 | 28
participants | 1 | 0
Statistical Analysis 1: Comparison: Ketamine vs Saline; Test type: Superiority or Other; p = 0.313, Chi-squared

26. Secondary Outcome: Allodynia as Detected With a Soft Brush in the Thenar Eminence Before the Procedure
Description: The evaluations using the soft brush were performed in the thenar eminence of the nondominant hand before the procedure
Time Frame: Before the procedure (Baseline)
Measure: Number; unit: participants
Arm/Group | Ketamine | Saline
Number analyzed (Participants) | 28 | 28
participants | 1 | 0
Statistical Analysis 1: Comparison: Ketamine vs Saline; Test type: Superiority or Other; p = 0.313, Chi-squared

27. Secondary Outcome: Allodynia as Detected With a Soft Brush in the Thenar Eminence 24 h After the Procedure
Description: The evaluations using the soft brush were performed in the thenar eminence of the non dominant hand 24 h after the procedure
Time Frame: 24 h after the procedure
Measure: Number; unit: participants
Arm/Group | Ketamine | Saline
Number analyzed (Participants) | 28 | 28
participants | 1 | 3
Statistical Analysis 1: Comparison: Ketamine vs Saline; Test type: Superiority or Other; p = 0.611, Chi-squared

28. Secondary Outcome: Serum Level of Interleukin (IL)-6 Before the Procedure
Description: Blood samples were drawn in ethylenediaminetetraacetic acid (EDTA) tubes before the surgery. The blood was centrifuged to separate the plasma and was stored at -70°C. IL-6 was analyzed using the enzyme-linked immunosorbent assay (ELISA) methodology.
Time Frame: Baseline (Before the procedure)
Measure: Mean (Standard Deviation); unit: picogram/milliliter
Arm/Group | Ketamine | Saline
Number analyzed (Participants) | 28 | 28
picogram/milliliter | 3.3 (9.5) | 2.1 (3.4)
Statistical Analysis 1: Comparison: Ketamine vs Saline; Test type: Superiority or Other; p = 0.312, t-test, 2 sided

29. Secondary Outcome: Serum Level of Interleukin (IL)-6 5 h After the Procedure
Description: Blood samples were drawn in ethylenediaminetetraacetic acid (EDTA) tubes 5 h after the surgery. The blood was centrifuged to separate the plasma and was stored at -70°C. IL-6 was analyzed using the enzyme-linked immunosorbent assay (ELISA) methodology.
Time Frame: 5 h after the procedure
Measure: Mean (Standard Deviation); unit: picogram/milliliter
Arm/Group | Ketamine | Saline
Number analyzed (Participants) | 28 | 28
picogram/milliliter | 29.3 (23.6) | 34.8 (48.7)
Statistical Analysis 1: Comparison: Ketamine vs Saline; Test type: Superiority or Other; p = 0.676, t-test, 2 sided

30. Secondary Outcome: Serum Level of Interleukin (IL)-6 24 h After the Procedure
Description: Blood samples were drawn in ethylenediaminetetraacetic acid (EDTA) tubes 24 h after the surgery. The blood was centrifuged to separate the plasma and was stored at -70°C. IL-6 was analyzed using the enzyme-linked immunosorbent assay (ELISA) methodology.
Time Frame: 24 h after the procedure
Measure: Mean (Standard Deviation); unit: picogram/milliliter
Arm/Group | Ketamine | Saline
Number analyzed (Participants) | 28 | 28
picogram/milliliter | 24.1 (21.3) | 24.8 (31.5)
Statistical Analysis 1: Comparison: Ketamine vs Saline; Test type: Superiority or Other; p = 0.938, t-test, 2 sided

31. Secondary Outcome: Serum Level of Interleukin (IL)-8 Before the Procedure
Description: Blood samples were drawn in ethylenediaminetetraacetic acid (EDTA) tubes before the surgery. The blood was centrifuged to separate the plasma and was stored at -70°C. IL-8 was analyzed using the enzyme-linked immunosorbent assay (ELISA) methodology.
Time Frame: Baseline (Before the procedure)
Measure: Mean (Standard Deviation); unit: picogram/milliliter
Arm/Group | Ketamine | Saline
Number analyzed (Participants) | 28 | 28
picogram/milliliter | 3.3 (4.1) | 2.2 (3.2)
Statistical Analysis 1: Comparison: Ketamine vs Saline; Test type: Superiority or Other; p = 0.385, t-test, 2 sided

32. Secondary Outcome: Serum Level of Interleukin (IL)-8 5 h After the Procedure
Description: Blood samples were drawn in ethylenediaminetetraacetic acid (EDTA) tubes 5 h after the surgery. The blood was centrifuged to separate the plasma and was stored at -70°C. IL-8 was analyzed using the enzyme-linked immunosorbent assay (ELISA) methodology.
Time Frame: 5 h after the procedure
Measure: Mean (Standard Deviation); unit: picogram/milliliter
Arm/Group | Ketamine | Saline
Number analyzed (Participants) | 28 | 28
picogram/milliliter | 8.0 (6.8) | 11.3 (15.1)
Statistical Analysis 1: Comparison: Ketamine vs Saline; Test type: Superiority or Other; p = 0.422, t-test, 2 sided

33. Secondary Outcome: Serum Level of Interleukin (IL)-8 24 h After the Procedure
Description: Blood samples were drawn in ethylenediaminetetraacetic acid (EDTA) tubes 24 h after the surgery. The blood was centrifuged to separate the plasma and was stored at -70°C. IL-8 was analyzed using the enzyme-linked immunosorbent assay (ELISA) methodology.
Time Frame: 24 h after the procedure
Measure: Mean (Standard Deviation); unit: picogram/milliliter
Arm/Group | Ketamine | Saline
Number analyzed (Participants) | 28 | 28
picogram/milliliter | 6.0 (7.2) | 4.5 (6.1)
Statistical Analysis 1: Comparison: Ketamine vs Saline; Test type: Superiority or Other; p = 0.500, t-test, 2 sided

34. Secondary Outcome: Serum Level of Interleukin (IL)-10 Before the Procedure
Description: as for outcome 28
Time Frame: Baseline (Before the procedure)
Measure: Mean (Standard Deviation); unit: picogram/milliliter
Arm/Group | Ketamine | Saline
Number analyzed (Participants) | 28 | 28
picogram/milliliter | 7.8 (20) | 1.9 (3.3)
Statistical Analysis 1: Comparison: Ketamine vs Saline; Test type: Superiority or Other; p = 0.435, t-test, 2 sided

35. Secondary Outcome: Serum Level of Interleukin (IL)-10 5h After the Procedure
Description: Blood samples were drawn in ethylenediaminetetraacetic acid (EDTA) tubes 5 h after the surgery. The blood was centrifuged to separate the plasma and was stored at -70°C. IL-10 was analyzed using the enzyme-linked immunosorbent assay (ELISA) methodology.
Time Frame: 5h after the procedure
Measure: Mean (Standard Deviation); unit: picogram/milliliter
Arm/Group | Ketamine | Saline
Number analyzed (Participants) | 28 | 28
picogram/milliliter | 9.1 (19.1) | 5.5 (7.9)
Statistical Analysis 1: Comparison: Ketamine vs Saline; Test type: Superiority or Other; p = 0.745, t-test, 2 sided

36. Secondary Outcome: Serum Level of Interleukin (IL)-10 24 h After the Procedure
Description: as for outcome 30
Time Frame: 24 h after the procedure
Measure: Mean (Standard Deviation); unit: picogram/milliliter
Arm/Group | Ketamine | Saline
Number analyzed (Participants) | 28 | 28
picogram/milliliter | 8.6 (18.5) | 5.0 (5.5)
Statistical Analysis 1: Comparison: Ketamine vs Saline; Test type: Superiority or Other; p = 0.557, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 24 hours
Groups:
- Ketamine: A cardioscope, a capnograph, a pulse oximeter, and a noninvasive blood pressure meter were used to monitor the patients. Propofol (2-4 mg/kg), 1 μg/kg remifentanil, and atracurium (0.5 mg/kg) were administered for intubation. Atracurium was titrated to maintain muscle relaxation. Anesthesia was maintained with remifentanil, 0.8% isoflurane, and 50% oxygen without nitrous oxide. Infusion of the solutions was continued until skin closure.
  The patients in group ketamine received remifentanil (0.4 μg/kg/min) and (ketamine 5 μg/kg/min). Remifentanil was administered as necessary until skin closure. Neostigmine was used for antagonizing the neuromuscular block.
Arm/Group | Ketamine | Saline
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 16/28 | 8/28
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ketamine (N=28) | Saline (N=28)
Vomiting (Gastrointestinal disorders) | 16 | 8
Diplopia/nystagmus (Eye disorders) | 5 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No